CLINICAL TRIAL: NCT02710487
Title: Awake & Move. Role of Nocturnal Sleep and Rapid Eye Movement Sleep at Morning Awakening on Sleep Benefit in Parkinson's Disease. An Interventional Cross-over Study.
Brief Title: Sleep, Awake & Move - Part II
Acronym: SA&M-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurocenter of Southern Switzerland (Other)
Collaborators: Parkinson Schweiz (Other); Ente Ospedaliero Cantonale, Bellinzona (Other); Penn State University (Other)
Responsible Party: Principal Investigator, Pietro Luca Ratti, MD, PhD, Neurocenter of Southern Switzerland
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: EOC.NSI.LS.15.3.II
Record Dates: First submitted 2016-03-12; First posted 2016-03-16 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease, Sleep Benefit
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Awakening from NREM vs. REM sleep.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The sleep technician in charge to apply the study intervention was the only person to be aware of the sleep phase the patient was awaken from.
Oversight: Data Monitoring Committee: No

ARMS (2):
- REM Sleep Awakening (REMSA) (Experimental): The investigators will actively awaken each subject from nocturnal REM sleep in a sleep laboratory setting, in the hour preceding her/his habitual wake time.
  Interventions: Behavioral: REMSA
- NREM Sleep Awakening (NREMSA) (Experimental): Awakening from the NREM sleep stage N2 will be the control intervention.
  Interventions: Behavioral: NREMSA

INTERVENTIONS:
Behavioral: REMSA — Awakening from REM sleep during the last hour of the sleep period
  Arms: REM Sleep Awakening (REMSA)
Behavioral: NREMSA — Awakening from N2 (NREM) sleep during the last hour of the sleep period
  Arms: NREM Sleep Awakening (NREMSA)

SUMMARY:
Sleep benefit (SB) is a prominent spontaneous, apparently unpredictable, transitory improvement in motor function reported by around 50% of patients affected by Parkinson's Disease (PD) after sleep and before taking their first dose of dopaminergic medications. The aim of this study is to test the hypothesis that objective and/or subjective improvement of motor function might be due to a carry-over effect of Rapid Eye Movements (REM) sleep at awakening from this sleep phase.

DETAILED DESCRIPTION:
The "Awake & Move" study is the second part of the Sleep, Awake & Move project. This study will be conducted in a subgroup of unselected, consecutive patients having completed the part I of the Sleep, Awake & Move project (i.e. the "Sleep & Move" study). The investigators plan to explore the carry-over effect of REM sleep on motor function in a subgroup of PD subjects p. In this interventional study the investigators expect to induce SB by awakening the subjects from nocturnal REM sleep in a sleep laboratory setting, but not from Non-Rapid Eye Movements (NREM) sleep (control intervention).

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria of idiopathic Parkinson's disease (UKPDBB)
* Mild to moderate disease (Hoehn & Yahr score ≥ 1 and < 3)
* Mentally and physically capable to give informed consent
* Stable antiparkinsonian and psychotropic therapy for the last 30 days

Exclusion Criteria:

* Atypical parkinsonian syndrome
* Cognitive impairment (MMSE ≥ 26)
* Deep brain stimulation
* History of cerebro-vascular disease, epilepsy, or other disabling neurological diseases
* Psychiatric disorders, excepting mild depression
* Alcohol abuse
* Other clinically significant severe concomitant disease states
* Inability to follow the procedures of the study (e.g. due to language problems, psychological disorders, etc.)
* Participation in another study with investigational drug within the 60 days preceding and during the present project.
* subjects with (a) sleep-disordered breathing [Respiratory Disorder Index (RDI)≥ 5] and (b) with no clear-cut distinction of REM and NREM sleep, based on a video-polysomongraphical recording.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Overnight change in objective motor performance | 12 hours
  The change of objective measures of morning motor performance at awakening from REM sleep compared to the morning motor performance at awakening from NREM sleep (stage N2), within the same subjects, by mean of an electronic finger tapping test and the Movement Disorders Society Unified Parkinson's Disease Rating Scale motor examination (MDS-UPDRS-III).

SECONDARY OUTCOMES:
Overnight change in subjective motor performance | 12 hours
  The change of subjective measures of morning motor performance at awakening from REM sleep compared to the morning motor performance at awakening from NREM sleep (stage N2), within the same subjects, by mean of the Scale for Outcome in Parkinson's Disease Diary Card (SCOPA-DC) and a visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Luca Ratti, MD, PhD, Principal Investigator — Neurocenter of Southern Switzerland
Locations (1):
- Sleep and Epilepsy center Department of Neurology, Neurocenter of Southern Switzerland, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Cock VC, Vidailhet M, Leu S, Texeira A, Apartis E, Elbaz A, Roze E, Willer JC, Derenne JP, Agid Y, Arnulf I. Restoration of normal motor control in Parkinson's disease during REM sleep. Brain. 2007 Feb;130(Pt 2):450-6. doi: 10.1093/brain/awl363. PMID 17235126
- [Background] Stefani A, Galati S, Peppe A, Bassi A, Pierantozzi M, Hainsworth AH, Bernardi G, Orlacchio A, Stanzione P, Mazzone P. Spontaneous sleep modulates the firing pattern of parkinsonian subthalamic nucleus. Exp Brain Res. 2006 Jan;168(1-2):277-80. doi: 10.1007/s00221-005-0175-y. Epub 2005 Nov 18. PMID 16328297
- [Background] Urrestarazu E, Iriarte J, Alegre M, Clavero P, Rodriguez-Oroz MC, Guridi J, Obeso JA, Artieda J. Beta activity in the subthalamic nucleus during sleep in patients with Parkinson's disease. Mov Disord. 2009 Jan 30;24(2):254-60. doi: 10.1002/mds.22351. PMID 18951542
- [Background] van Gilst MM, Bloem BR, Overeem S. "Sleep benefit" in Parkinson's disease: a systematic review. Parkinsonism Relat Disord. 2013 Jul;19(7):654-9. doi: 10.1016/j.parkreldis.2013.03.014. Epub 2013 Apr 21. PMID 23615667
- [Background] Merello M, Hughes A, Colosimo C, Hoffman M, Starkstein S, Leiguarda R. Sleep benefit in Parkinson's disease. Mov Disord. 1997 Jul;12(4):506-8. doi: 10.1002/mds.870120405. PMID 9251067
- [Background] Currie LJ, Bennett JP Jr, Harrison MB, Trugman JM, Wooten GF. Clinical correlates of sleep benefit in Parkinson's disease. Neurology. 1997 Apr;48(4):1115-7. doi: 10.1212/wnl.48.4.1115. PMID 9109914
- [Background] Tandberg E, Larsen JP, Karlsen K. Excessive daytime sleepiness and sleep benefit in Parkinson's disease: a community-based study. Mov Disord. 1999 Nov;14(6):922-7. doi: 10.1002/1531-8257(199911)14:63.0.co;2-7. PMID 10584665
- [Background] Bateman DE, Levett K, Marsden CD. Sleep benefit in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1999 Sep;67(3):384-5. doi: 10.1136/jnnp.67.3.384. No abstract available. PMID 10449564
- [Background] Sherif E, Valko PO, Overeem S, Baumann CR. Sleep benefit in Parkinson's disease is associated with short sleep times. Parkinsonism Relat Disord. 2014 Jan;20(1):116-8. doi: 10.1016/j.parkreldis.2013.09.005. Epub 2013 Sep 12. PMID 24084381
- [Background] Hogl BE, Gomez-Arevalo G, Garcia S, Scipioni O, Rubio M, Blanco M, Gershanik OS. A clinical, pharmacologic, and polysomnographic study of sleep benefit in Parkinson's disease. Neurology. 1998 May;50(5):1332-9. doi: 10.1212/wnl.50.5.1332. PMID 9595983
- [Background] Hogl B, Peralta C, Wetter TC, Gershanik O, Trenkwalder C. Effect of sleep deprivation on motor performance in patients with Parkinson's disease. Mov Disord. 2001 Jul;16(4):616-21. doi: 10.1002/mds.1138. PMID 11481684
- [Background] Hogl B, Gershanik O. Sleep benefit in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2000 Jun;68(6):798-9. doi: 10.1136/jnnp.68.6.798a. No abstract available. PMID 10877630
- [Background] Factor SA, Weiner WJ. 'Sleep benefit' in Parkinson's disease. Neurology. 1998 May;50(5):1514-5. doi: 10.1212/wnl.50.5.1514-b. No abstract available. PMID 9596032
- [Background] Noyce AJ, Nagy A, Acharya S, Hadavi S, Bestwick JP, Fearnley J, Lees AJ, Giovannoni G. Bradykinesia-akinesia incoordination test: validating an online keyboard test of upper limb function. PLoS One. 2014 Apr 29;9(4):e96260. doi: 10.1371/journal.pone.0096260. eCollection 2014. PMID 24781810